CLINICAL TRIAL: NCT05163522
Title: A Randomized, Double-Blind (Sponsor Unblinded), Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Orally Administered VH4004280 in Healthy Participants
Brief Title: First-Time-in-Human (FTIH) Study to Evaluate the Safety, Tolerability and Pharmacokinetics (PK) of VH4004280 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 217058
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: First-time-in-human; GSK4004280; VH4004280; HIV-1 capsid inhibitor; Single ascending doses; Multiple ascending doses
MeSH Terms: conditions — HIV Infections | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind (sponsor unblinded) study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) (Placebo Comparator): Healthy participants were given a single oral dose of placebo on Day 1 and were followed up to approximately Day 49.
  Interventions: Drug: Placebo
- Part 1 (SAD): VH4004280 10 mg PiB (Experimental): Healthy participants were given a single oral dose of 10 mg VH4004280 PiB on Day 1 and were followed up to approximately Day 49.
  Interventions: Drug: VH4004280
- Part 1 (SAD): VH4004280 50 mg PiB (Experimental): Healthy participants were given a single oral dose of 50 mg VH4004280 PiB on Day 1 and were followed up to approximately Day 49.
  Interventions: Drug: VH4004280
- Part 1 (SAD): VH4004280 150 mg PiB (Experimental): Healthy participants were given a single oral dose of 150 mg VH4004280 PiB on Day 1 and were followed up to approximately Day 49.
  Interventions: Drug: VH4004280
- Part 1 (SAD): VH4004280 450 mg PiB (Experimental): Healthy participants were given a single oral dose of 450 mg VH4004280 PiB on Day 1 and were followed up to approximately Day 49.
  Interventions: Drug: VH4004280
- Part 1 (SAD): VH4004280 900 mg PiB (Experimental): Healthy participants were given a single oral dose of 900 mg VH4004280 PiB on Day 1 and were followed up to approximately Day 49.
  Interventions: Drug: VH4004280
- Part 2 Multiple Ascending Dose (MAD): Placebo PiB (Placebo Comparator): Healthy participants were given a dose of placebo once daily (QD) for a 14-day period and were followed up to approximately Day 63.
  Interventions: Drug: Placebo
- Part 2 (MAD): VH4004280 100 mg PiB (Experimental): Healthy participants were given a dose of 100 mg VH4004280 PiB QD for a 14-day period and were followed up to approximately Day 63.
  Interventions: Drug: VH4004280
- Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB (Experimental): Healthy participants were given a dose of 250 mg VH4004280 PiB QD for a 14-day period, and a single dose of Midazolam on days 1, 2, and 15, and were followed up to approximately Day 63.
  Interventions: Drug: VH4004280; Drug: Midazolam
- Part 2 (MAD): VH4004280 350 mg PiB (Experimental): Healthy participants were given a dose of 350 mg VH4004280 PiB QD for a 14-day period and were followed up to approximately Day 63.
  Interventions: Drug: VH4004280
- Part 3 (Single dose): VH4004280 450 mg tablet (Experimental): Healthy participants were given a single oral dose of VH4004280 450 mg tablet at Day 1 and were followed up to approximately Day 49.
  Interventions: Drug: VH4004280

INTERVENTIONS:
Drug: VH4004280 — VH4004280 will be administered.
  Other Names: GSK4004280
  Arms: Part 1 (SAD): VH4004280 10 mg PiB; Part 1 (SAD): VH4004280 150 mg PiB; Part 1 (SAD): VH4004280 450 mg PiB; Part 1 (SAD): VH4004280 50 mg PiB; Part 1 (SAD): VH4004280 900 mg PiB; Part 2 (MAD): VH4004280 100 mg PiB; Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB; Part 2 (MAD): VH4004280 350 mg PiB; Part 3 (Single dose): VH4004280 450 mg tablet
Drug: Placebo — Placebo will be administered.
  Arms: Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB); Part 2 Multiple Ascending Dose (MAD): Placebo PiB
Drug: Midazolam — Midazolam will be administered
  Arms: Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB

SUMMARY:
This FTIH study aims to evaluate the safety, tolerability and PK of the novel investigational Human immunodeficiency virus (HIV)-1 capsid inhibitor VH4004280 in healthy adults. The study will be conducted in 3 parts: Part 1 will investigate single ascending doses (SAD), Part 2 will investigate multiple ascending doses and drug-drug interaction (MAD/MAD DDI) Part 3 will investigate single dose relative bioavailability (RBA) of a new formulation of VH4004280.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 to 55 years of age inclusive.
* Participants who are overtly healthy.
* Male or female participants of non-childbearing potential.
* Capable of giving signed informed consent.

Exclusion criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neurological or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study drug or interfering with the interpretation of data.
* Abnormal blood pressure.
* Symptomatic herpes zoster.
* Evidence of active or latent tuberculosis (TB).
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) greater than (>)450 milliseconds (msec).
* Past or intended use of over-the-counter or prescription medication including herbal medications.
* Live vaccine(s) within 1 month prior to screening or plans to receive such vaccines during the study.
* Exposure to more than 4 new investigational products within 12 months prior to the first dosing day.
* Current enrollment or past participation in another investigational study.
* ALT >1.5 times upper limit of normal (ULN), total bilirubin >1.5 times ULN, and/or estimated serum creatinine clearance less than 60 milliliters per minute.
* History of or current infection with hepatitis B or hepatitis C.
* Positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) test, having signs and symptoms, or having contact with known Coronavirus Disease-2019 (COVID-19) positive person/s.
* Positive HIV antibody test.
* User of tobacco or nicotine-containing products, regular alcohol consumption and/or regular use of known drugs of abuse.
* Sensitivity to the study drug, or components thereof.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf

REFERENCES:
- [Derived] Thakkar N, Griesel R, Pierce A, Bainbridge V, Shepherd B, Angelis K, Tomlinson A, Gandhi Y, Brimhall D, Anderson D, Andrews S, Acuipil C, McCoig C, Baker M, Benn P. Clinical Pharmacokinetics and Safety of a New HIV-1 Capsid Inhibitor, VH4004280, After Oral Administration in Adults Without HIV. Infect Dis Ther. 2025 Jun;14(6):1313-1326. doi: 10.1007/s40121-025-01154-x. Epub 2025 Apr 26. PMID 40287607

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB | Part 3 (Single Dose): VH4004280 450 mg Tablet
Started | 10 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB | Part 3 (Single Dose): VH4004280 450 mg Tablet | Total
Number analyzed (Participants) | 10 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 73
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 34.0 (7.21) | 33.8 (8.13) | 30.0 (9.36) | 31.5 (6.28) | 27.7 (6.44) | 31.5 (6.02) | 36.2 (7.68) | 33.5 (9.09) | 34.0 (10.74) | 42.3 (11.08) | 43.5 (7.06) | 34.27 (8.898)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 10 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 5 | 72
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 7
  Black or African American | 3 | 2 | 1 | 3 | 5 | 2 | 2 | 4 | 6 | 3 | 3 | 34
  Native Hawaiian or other Pacific Islander | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 4 | 2 | 5 | 3 | 1 | 4 | 4 | 0 | 1 | 3 | 1 | 28
  Multiple | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Any Adverse Events (AEs) and by Severity
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a study intervention whether or not considered related to the study intervention. The Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric AE was used for all AE severity grading, where Grade 1=Mild symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated, 2=Moderate symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated, 3=Severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated, 4=Potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability or death, 5=Death.
Time Frame: Up to Day 49
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 1 (SAD) who received 1 full dose of study treatment. The participants were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 10 | 6 | 7 | 6 | 6 | 6
Participants
  Any AEs | 4 | 2 | 3 | 0 | 0 | 1
  Grade 1 AEs | 3 | 2 | 3 | 0 | 0 | 1
  Grade 2 AEs | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 AEs | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 AEs | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 AEs | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2: Number of Participants With Any AEs and by Severity
Description: The DAIDS Table for Grading the Severity of Adult and Pediatric AE was used for all AE severity grading, where Grade 1=Mild symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated, 2=Moderate symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated, 3=Severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated, 4=Potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability or death, 5=Death.
Time Frame: Up to Day 63
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 2 (MAD) who received at least 1 full or partial dose of study treatment. The participants were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 6 | 8 | 6
Participants
  Any AEs | 3 | 4 | 7 | 4
  Grade 1 AEs | 3 | 4 | 4 | 2
  Grade 2 AEs | 0 | 0 | 3 | 0
  Grade 3 AEs | 0 | 0 | 0 | 1
  Grade 4 AEs | 0 | 0 | 0 | 1
  Grade 5 AEs | 0 | 0 | 0 | 0

3. Primary Outcome: Part 3: Number of Participants With Any AEs and by Severity
Description: as for outcome 2
Time Frame: Up to Day 49
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 3 (Single Dose) who received 1 single dose of study treatment. The participants were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 (Single Dose): VH4004280 450 mg Tablet
Number analyzed (Participants) | 6
Participants
  Any AEs | 3
  Grade 1 AEs | 2
  Grade 2 AEs | 0
  Grade 3 AEs | 1
  Grade 4 AEs | 0
  Grade 5 AEs | 0

4. Primary Outcome: Part 2: Number of Participants Discontinuing Treatment Due to AEs
Description: Number of participants who discontinued treatment due to AEs are presented.
Time Frame: Up to Day 63
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 6 | 8 | 6
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Part 1: Absolute Values of Liver Panel Parameters: Direct Bilirubin and Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of bilirubin. Standard Deviation (SD)=0.0000 is defined as following: if all participants analyzed for a specific parameter at a specific time point have the same value, then SD is equal with 0.0000.
Time Frame: Up to Day 49
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 1 (SAD) who received 1 full dose of study treatment. The participants were analyzed according to the treatment they actually received. Only those participants with data available at specified time points were analyzed for the specific category titles.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (μmol/L)
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 10 | 6 | 7 | 6 | 6 | 6
Micromoles per liter (μmol/L)
  Direct Bilirubin, Baseline (Day 1) | 2.5650 (1.20915) | 1.9950 (0.69810) | 2.9314 (0.83439) | 2.2800 (1.39621) | 2.2800 (0.88304) | 2.8500 (0.88304)
  Direct Bilirubin, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  Direct Bilirubin, Day 2 | 2.7170 (1.24620) | 2.5080 (0.59891) | 2.9559 (1.17113) | 2.0520 (1.03734) | 2.7360 (0.93661) | 3.0780 (1.27507)
  Direct Bilirubin, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 3 | 2.7018 (1.15078) | 2.4795 (0.51584) | 2.7075 (0.98776) | 1.8525 (1.07834) | 2.3655 (0.87472) | 3.0495 (1.23033)
  Direct Bilirubin, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  Direct Bilirubin, Day 4 | 2.4966 (1.36847) | 2.0235 (0.79043) | 2.7360 (0.87193) | 1.9836 (0.73151) | 2.2515 (1.11566) | 2.6790 (1.02410)
  Direct Bilirubin, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 5 | 2.7360 (1.18198) | 2.6505 (0.63753) | 2.5080 (0.73085) | 1.9665 (0.81472) | 2.8215 (0.75512) | 2.8215 (0.98381)
  Direct Bilirubin, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 6 | 2.5650 (0.68400) | 2.6505 (0.69038) | 2.3085 (0.77045) | 1.7955 (0.89673) | 2.3655 (0.98182) | 2.8785 (1.17190)
  Direct Bilirubin, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 7 | 2.8899 (1.24216) | 2.4795 (0.63753) | 2.2800 (0.70643) | 1.9095 (0.75253) | 2.3370 (1.26894) | 2.5935 (0.95770)
  Direct Bilirubin, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  Direct Bilirubin, Day 14 | 2.3598 (0.77234) | 1.7100 (0.00000) | 1.5732 (0.37072) | 1.6245 (0.86351) | 2.2230 (0.29618) | 2.6790 (1.60291)
  Direct Bilirubin, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 21 | 2.5308 (1.19238) | 2.1375 (0.95974) | 2.3085 (0.94747) | 1.4250 (0.49166) | 2.4795 (0.83598) | 2.0520 (0.98529)
  Direct Bilirubin, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Direct Bilirubin, Day 28 | 2.8215 (1.67400) | 2.0805 (0.97585) | 2.3256 (0.81651) | 1.6530 (0.51490) | 3.2490 (1.34646) | 2.3370 (0.88304)
  Direct Bilirubin, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  Direct Bilirubin, Day 35 | 2.3598 (1.25348) | 2.1090 (0.69810) | 2.2800 (0.91556) | 1.7385 (0.83364) | 2.2800 (1.00682) | 1.9494 (0.76090)
  Direct Bilirubin, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Direct Bilirubin, Day 42 | 2.9355 (2.10105) |  |  | 1.6530 (0.69810) | 2.7360 (1.38499) | 2.7645 (1.44053)
  Direct Bilirubin, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Direct Bilirubin, Day 49 | 2.9355 (1.48452) |  |  | 1.5675 (0.58657) | 2.6505 (1.15852) | 2.6505 (1.49759)
  Total Bilirubin, Baseline (Day 1) | 13.1670 (6.84237) | 12.5400 (3.84908) | 14.9014 (3.65613) | 12.2550 (8.47558) | 11.6850 (5.00498) | 10.8300 (5.26132)
  Total Bilirubin, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  Total Bilirubin, Day 2 | 14.8770 (7.69405) | 11.9130 (3.49052) | 13.4357 (4.91245) | 10.7730 (6.63074) | 17.9835 (7.41865) | 16.2735 (7.49161)
  Total Bilirubin, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 3 | 14.2956 (6.79530) | 11.7705 (3.38635) | 12.1410 (4.37573) | 10.4595 (7.28983) | 15.5040 (7.42594) | 15.5895 (6.56018)
  Total Bilirubin, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 5
  Total Bilirubin, Day 4 | 13.6287 (8.26482) | 9.4620 (3.81091) | 14.2215 (6.54322) | 10.6704 (7.32172) | 15.8460 (5.98125) | 13.5090 (6.44718)
  Total Bilirubin, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 5 | 13.5603 (6.89113) | 11.6565 (3.15571) | 11.8275 (4.79461) | 10.6875 (5.85984) | 15.7320 (7.04470) | 14.7345 (5.17813)
  Total Bilirubin, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 6 | 12.9618 (4.88926) | 12.1125 (3.92990) | 9.6330 (3.97319) | 9.3480 (6.12902) | 13.9365 (7.53701) | 14.3640 (5.24388)
  Total Bilirubin, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 7 | 13.8510 (7.21180) | 10.6020 (3.25350) | 9.9465 (2.53730) | 10.7160 (5.72854) | 16.6725 (8.20640) | 12.5400 (4.43239)
  Total Bilirubin, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  Total Bilirubin, Day 14 | 10.4139 (2.46942) | 6.7545 (3.25125) | 7.2846 (2.33087) | 7.9515 (4.34050) | 11.1150 (0.91289) | 11.7990 (7.42857)
  Total Bilirubin, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 21 | 12.4317 (5.82742) | 9.6045 (5.04078) | 10.2885 (3.37424) | 7.5525 (3.38980) | 12.4830 (4.36636) | 8.9205 (3.94920)
  Total Bilirubin, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Total Bilirubin, Day 28 | 13.1670 (9.01537) | 9.1200 (4.86394) | 10.1916 (4.40238) | 7.9800 (2.95720) | 16.7580 (9.74550) | 11.4000 (3.21674)
  Total Bilirubin, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  Total Bilirubin, Day 35 | 12.0042 (7.37960) | 8.5785 (3.90002) | 10.0605 (3.87143) | 8.4360 (4.45476) | 11.3715 (7.28046) | 8.7552 (2.95786)
  Total Bilirubin, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Total Bilirubin, Day 42 | 14.8485 (12.01166) |  |  | 8.2080 (4.29070) | 15.5895 (10.02324) | 12.9675 (6.50917)
  Total Bilirubin, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Total Bilirubin, Day 49 | 14.0505 (7.95429) |  |  | 8.8350 (3.94512) | 14.8200 (6.47967) | 12.7680 (8.27588)

6. Primary Outcome: Part 1: Absolute Values of Liver Panel Parameters: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of ALP, ALT and AST.
Time Frame: Up to Day 49
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 10 | 6 | 7 | 6 | 6 | 6
International units per liter (IU/L)
  ALP, Baseline (Day 1) | 51.8 (9.39) | 64.7 (10.88) | 67.1 (27.91) | 69.0 (25.04) | 64.0 (11.10) | 61.8 (15.41)
  ALP, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  ALP, Day 2 | 48.6 (7.52) | 59.0 (10.86) | 60.4 (23.56) | 63.5 (21.68) | 58.2 (10.61) | 54.5 (9.73)
  ALP, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 3 | 48.2 (4.57) | 58.8 (11.20) | 56.2 (21.44) | 63.0 (21.25) | 55.8 (10.76) | 52.5 (10.29)
  ALP, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  ALP, Day 4 | 49.3 (6.60) | 60.5 (12.08) | 60.5 (19.36) | 58.6 (18.84) | 63.2 (10.57) | 52.8 (11.86)
  ALP, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 5 | 48.1 (8.16) | 59.2 (10.32) | 54.7 (20.65) | 63.3 (21.16) | 60.5 (9.57) | 57.7 (9.16)
  ALP, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 6 | 48.8 (6.44) | 62.5 (10.99) | 56.3 (21.10) | 63.0 (19.15) | 62.3 (10.01) | 54.5 (7.40)
  ALP, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 7 | 51.7 (7.30) | 64.3 (13.60) | 61.7 (17.18) | 64.3 (20.25) | 66.3 (11.41) | 56.8 (7.44)
  ALP, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  ALP, Day 14 | 54.8 (11.85) | 62.2 (6.97) | 59.6 (19.49) | 65.0 (21.48) | 66.4 (12.72) | 61.3 (8.62)
  ALP, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 21 | 53.0 (11.18) | 58.7 (9.50) | 62.2 (29.88) | 66.0 (22.33) | 61.5 (12.05) | 59.2 (8.70)
  ALP, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  ALP, Day 28 | 53.9 (12.35) | 57.5 (7.97) | 66.2 (43.85) | 65.5 (22.95) | 63.5 (10.82) | 65.5 (11.33)
  ALP, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  ALP, Day 35 | 52.9 (8.69) | 66.3 (12.80) | 62.3 (28.22) | 63.8 (23.56) | 64.7 (9.14) | 62.8 (8.07)
  ALP, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  ALP, Day 42 | 53.7 (9.75) |  |  | 63.3 (25.31) | 66.2 (9.54) | 63.2 (9.79)
  ALP, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  ALP, Day 49 | 54.3 (7.53) |  |  | 67.2 (27.21) | 66.7 (11.50) | 59.7 (6.41)
  ALT, Baseline (Day 1) | 18.4 (5.60) | 22.8 (11.72) | 15.1 (4.85) | 20.7 (8.07) | 14.8 (2.93) | 16.0 (4.34)
  ALT, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  ALT, Day 2 | 18.3 (7.78) | 22.0 (16.60) | 15.6 (5.47) | 21.3 (9.61) | 15.7 (3.61) | 15.3 (3.08)
  ALT, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 3 | 18.6 (7.15) | 22.2 (17.23) | 15.8 (7.65) | 20.7 (9.09) | 15.8 (3.60) | 16.0 (4.52)
  ALT, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  ALT, Day 4 | 19.2 (6.60) | 23.2 (17.47) | 16.7 (8.94) | 22.4 (12.52) | 14.3 (3.20) | 16.2 (4.12)
  ALT, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 5 | 18.1 (6.30) | 21.7 (16.74) | 17.0 (10.84) | 24.5 (13.77) | 15.0 (2.68) | 16.0 (4.77)
  ALT, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 6 | 18.9 (7.96) | 22.5 (16.15) | 18.0 (12.98) | 24.2 (13.27) | 14.5 (3.02) | 18.8 (7.96)
  ALT, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 7 | 19.9 (9.97) | 23.5 (15.59) | 18.2 (12.83) | 24.7 (14.90) | 15.3 (3.20) | 20.8 (10.28)
  ALT, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  ALT, Day 14 | 26.1 (21.07) | 27.3 (17.90) | 18.0 (8.86) | 29.8 (21.29) | 22.0 (11.51) | 22.7 (13.87)
  ALT, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 21 | 23.4 (15.94) | 23.5 (13.98) | 20.2 (10.61) | 24.5 (10.54) | 19.2 (7.41) | 22.2 (15.66)
  ALT, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  ALT, Day 28 | 20.1 (10.02) | 33.7 (22.25) | 17.6 (8.50) | 24.2 (9.50) | 16.8 (6.37) | 20.8 (10.63)
  ALT, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  ALT, Day 35 | 19.8 (10.78) | 28.5 (15.42) | 17.8 (8.35) | 23.5 (5.75) | 21.3 (15.71) | 16.8 (3.70)
  ALT, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  ALT, Day 42 | 14.2 (3.60) |  |  | 25.5 (6.02) | 16.3 (4.23) | 17.5 (4.76)
  ALT, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  ALT, Day 49 | 15.0 (4.34) |  |  | 27.8 (9.85) | 18.7 (10.23) | 17.2 (5.23)
  AST, Baseline (Day 1) | 17.3 (5.03) | 17.3 (5.82) | 15.1 (4.14) | 17.5 (3.62) | 15.0 (3.03) | 16.5 (3.51)
  AST, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  AST, Day 2 | 17.3 (7.97) | 16.3 (8.31) | 14.3 (3.40) | 16.5 (3.78) | 15.0 (2.97) | 15.8 (2.71)
  AST, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 3 | 16.4 (4.33) | 16.0 (7.56) | 14.8 (4.07) | 16.7 (3.44) | 14.7 (2.80) | 15.2 (2.14)
  AST, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  AST, Day 4 | 15.8 (3.82) | 16.7 (7.76) | 15.3 (3.83) | 18.4 (5.46) | 13.3 (2.42) | 15.5 (2.81)
  AST, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 5 | 14.8 (2.90) | 14.8 (6.34) | 14.8 (3.92) | 18.5 (5.05) | 13.7 (1.63) | 15.8 (2.14)
  AST, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 6 | 15.6 (3.13) | 16.0 (6.42) | 15.7 (5.43) | 17.7 (5.57) | 14.3 (1.21) | 16.7 (2.34)
  AST, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 7 | 16.5 (3.84) | 16.8 (5.38) | 15.8 (4.36) | 18.2 (5.49) | 15.3 (2.16) | 18.0 (3.10)
  AST, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  AST, Day 14 | 40.0 (71.85) | 18.0 (6.13) | 14.2 (5.22) | 20.7 (7.81) | 20.0 (7.97) | 17.5 (3.62)
  AST, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 21 | 17.9 (6.82) | 18.7 (5.28) | 18.3 (8.09) | 19.5 (3.78) | 17.3 (2.94) | 18.2 (5.38)
  AST, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  AST, Day 28 | 16.8 (3.39) | 23.0 (6.54) | 17.0 (6.04) | 20.3 (4.08) | 16.3 (1.75) | 16.8 (1.94)
  AST, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  AST, Day 35 | 17.4 (4.70) | 20.5 (6.19) | 18.3 (7.50) | 21.7 (4.50) | 18.5 (4.32) | 18.0 (2.65)
  AST, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  AST, Day 42 | 14.8 (1.72) |  |  | 22.8 (2.99) | 16.3 (2.58) | 16.8 (3.19)
  AST, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  AST, Day 49 | 15.2 (2.04) |  |  | 23.3 (6.15) | 18.2 (2.93) | 18.0 (5.22)

7. Primary Outcome: Part 2: Absolute Values of Liver Panel Parameters: Direct Bilirubin and Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of bilirubin. Standard Deviation (SD)=0.00000 is defined as following: if all participants analyzed for a specific parameter at a specific time point have the same value, then SD is equal with 0.00000.
Time Frame: Up to Day 63
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 2 (MAD) who received at least 1 full or partial dose of study treatment. The participants were analyzed according to the treatment they actually received. Only those participants with data available at specified time points were analyzed for the specific category titles.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 6 | 8 | 6
μmol/L
  Direct Bilirubin, Baseline (Day 1) | 2.2800 (0.88304) | 2.8500 (1.39621) | 2.1375 (0.79158) | 1.7100 (0.00000)
  Direct Bilirubin, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 2 | 2.1803 (0.47090) | 3.1065 (1.34826) |  | 2.1375 (0.40103)
  Direct Bilirubin, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 3 | 2.2230 (0.24183) |  | 2.1589 (0.78595) |
  Direct Bilirubin, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 5 | 2.0948 (0.35253) | 3.1635 (1.82498) |  | 2.1945 (0.54524)
  Direct Bilirubin, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 6 | 2.2230 (0.00000) |  | 2.3940 (0.99289) |
  Direct Bilirubin, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 7 | 1.8383 (0.37917) | 2.9070 (1.75056) |  | 2.5650 (0.47141)
  Direct Bilirubin, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 8 | 2.3940 (0.72549) |  | 2.4795 (0.83272) |
  Direct Bilirubin, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  Direct Bilirubin, Day 11 | 2.2230 (0.72549) | 2.6505 (1.04948) |  | 2.4795 (0.58989)
  Direct Bilirubin, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 12 | 1.9665 (0.60458) |  | 2.5436 (0.76712) |
  Direct Bilirubin, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 14 | 1.5818 (0.29204) | 2.6220 (1.07426) |  | 1.9950 (0.33625)
  Direct Bilirubin, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 15 | 2.7360 (0.24183) |  | 2.8856 (0.78329) |
  Direct Bilirubin, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 21 | 1.7100 (0.46307) | 2.7360 (1.17978) |  | 2.5935 (0.34905)
  Direct Bilirubin, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 22 | 3.5055 (0.12092) |  | 3.2276 (0.93409) |
  Direct Bilirubin, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  Direct Bilirubin, Day 28 | 1.5732 (0.44262) | 2.0235 (0.64362) | 2.0948 (0.61145) | 1.8810 (0.49561)
  Direct Bilirubin, Day 35 | 1.7955 (0.28098) | 1.8810 (0.63982) | 2.1375 (0.59937) | 1.7955 (0.41536)
  Direct Bilirubin, Day 42 | 2.0520 (0.58241) | 2.0805 (0.77549) | 2.0306 (0.57401) | 1.5960 (0.35322)
  Direct Bilirubin, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  Direct Bilirubin, Day 49 | 2.1204 (0.66887) | 2.2230 (0.80206) | 2.2016 (0.59544) | 1.9095 (0.59646)
  Direct Bilirubin, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  Direct Bilirubin, Day 56 | 1.9095 (0.47656) | 2.2914 (1.08555) | 1.8810 (0.51706) | 1.7955 (0.49265)
  Direct Bilirubin, Day 63 | 1.7670 (0.38491) | 1.9095 (0.69601) | 1.8596 (0.83990) | 1.9665 (0.51584)
  Total Bilirubin, Baseline (Day 1) | 11.9700 (3.42000) | 15.1050 (6.87553) | 9.6188 (3.53265) | 8.2650 (1.28724)
  Total Bilirubin, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 2 | 10.6020 (2.39807) | 17.9550 (8.54521) |  | 11.6565 (2.67858)
  Total Bilirubin, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 3 | 16.3305 (6.40851) |  | 12.2051 (3.59151) |
  Total Bilirubin, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 5 | 10.6020 (2.08498) | 18.8670 (10.05775) |  | 13.0815 (4.18409)
  Total Bilirubin, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 6 | 15.1335 (4.71570) |  | 13.2525 (4.38546) |
  Total Bilirubin, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 7 | 9.0203 (1.14604) | 16.5015 (9.02436) |  | 14.8770 (3.05894)
  Total Bilirubin, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 8 | 16.5870 (8.94773) |  | 14.4281 (3.99249) |
  Total Bilirubin, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  Total Bilirubin, Day 11 | 9.4050 (3.62746) | 15.2190 (5.69715) |  | 13.0530 (2.43917)
  Total Bilirubin, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 12 | 11.4570 (0.72549) |  | 15.6893 (3.63062) |
  Total Bilirubin, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 14 | 7.3958 (1.36354) | 14.2500 (4.70504) |  | 13.9650 (2.37109)
  Total Bilirubin, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 15 | 15.5610 (4.11112) |  | 14.9839 (4.61559) |
  Total Bilirubin, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 21 | 7.6095 (1.74666) | 15.8175 (5.32110) |  | 14.9625 (2.61076)
  Total Bilirubin, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 22 | 19.9215 (5.92485) |  | 18.0833 (4.97435) |
  Total Bilirubin, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  Total Bilirubin, Day 28 | 8.3106 (2.41710) | 10.3170 (3.52221) | 9.7256 (2.84298) | 9.7755 (2.53499)
  Total Bilirubin, Day 35 | 9.2910 (1.47365) | 10.7730 (3.04361) | 10.3028 (2.29739) | 9.1200 (1.86591)
  Total Bilirubin, Day 42 | 10.6305 (4.12024) | 10.7445 (3.45304) | 10.2173 (3.00208) | 8.8920 (3.09505)
  Total Bilirubin, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  Total Bilirubin, Day 49 | 11.5254 (4.75214) | 12.1410 (3.91885) | 11.1791 (2.73896) | 9.7755 (3.40872)
  Total Bilirubin, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  Total Bilirubin, Day 56 | 10.1175 (5.17248) | 11.0466 (4.41233) | 8.3149 (1.86413) | 8.8065 (2.41770)
  Total Bilirubin, Day 63 | 8.9205 (2.27993) | 10.3455 (3.58815) | 8.9775 (3.69817) | 10.1745 (2.83829)

8. Primary Outcome: Part 2: Absolute Values of Liver Panel Parameters: ALP, ALT and AST
Description: as for outcome 6
Time Frame: Up to Day 63
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 6 | 8 | 6
IU/L
  ALP, Baseline (Day 1) | 66.2 (16.75) | 53.7 (10.01) | 57.5 (21.37) | 56.7 (11.41)
  ALP, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 2 | 69.0 (27.47) | 52.0 (8.97) |  | 56.2 (10.23)
  ALP, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 3 | 68.0 (5.66) |  | 58.4 (20.88) |
  ALP, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 5 | 64.3 (23.14) | 49.8 (6.79) |  | 57.2 (9.60)
  ALP, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 6 | 64.0 (4.24) |  | 55.6 (19.78) |
  ALP, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 7 | 64.8 (25.16) | 48.8 (7.39) |  | 56.5 (7.12)
  ALP, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 8 | 68.5 (9.19) |  | 55.8 (18.98) |
  ALP, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  ALP, Day 11 | 72.0 (2.83) | 47.5 (4.20) |  | 54.3 (11.47)
  ALP, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 12 | 71.0 (4.24) |  | 58.3 (21.97) |
  ALP, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 14 | 69.5 (24.52) | 47.7 (7.53) |  | 58.0 (12.20)
  ALP, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 15 | 66.0 (5.66) |  | 58.0 (19.09) |
  ALP, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 21 | 62.0 (19.41) | 50.5 (5.21) |  | 57.5 (11.64)
  ALP, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 22 | 70.5 (4.95) |  | 62.6 (19.53) |
  ALP, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALP, Day 28 | 61.4 (15.98) | 49.2 (11.69) | 59.8 (19.20) | 59.5 (10.73)
  ALP, Day 35 | 64.2 (17.88) | 53.0 (15.26) | 59.9 (17.10) | 53.0 (11.56)
  ALP, Day 42 | 67.7 (19.31) | 51.3 (11.76) | 62.1 (19.58) | 57.7 (12.09)
  ALP, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALP, Day 49 | 64.2 (16.81) | 51.0 (12.36) | 58.8 (18.48) | 54.0 (12.71)
  ALP, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  ALP, Day 56 | 69.0 (19.71) | 51.6 (11.15) | 62.8 (20.42) | 56.5 (7.20)
  ALP, Day 63 | 66.5 (17.44) | 53.8 (11.75) | 58.8 (18.97) | 57.3 (11.08)
  ALT, Baseline (Day 1) | 18.7 (11.98) | 19.0 (6.93) | 16.3 (5.04) | 19.5 (7.69)
  ALT, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 2 | 16.0 (9.42) | 19.2 (5.12) |  | 19.8 (7.65)
  ALT, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 3 | 19.0 (8.49) |  | 18.3 (4.43) |
  ALT, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 5 | 19.0 (8.76) | 19.5 (5.32) |  | 16.7 (6.28)
  ALT, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 6 | 15.0 (5.66) |  | 18.3 (5.26) |
  ALT, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 7 | 22.3 (12.50) | 24.7 (9.14) |  | 16.5 (6.47)
  ALT, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 8 | 15.0 (7.07) |  | 16.8 (5.39) |
  ALT, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  ALT, Day 11 | 21.0 (11.31) | 20.8 (3.86) |  | 14.8 (5.34)
  ALT, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 12 | 19.0 (8.49) |  | 19.1 (8.81) |
  ALT, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 14 | 33.3 (31.36) | 29.5 (14.01) |  | 16.7 (6.77)
  ALT, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 15 | 20.0 (7.07) |  | 21.5 (10.04) |
  ALT, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 21 | 24.5 (11.39) | 32.8 (15.35) |  | 23.2 (9.28)
  ALT, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 22 | 21.5 (3.54) |  | 24.1 (8.46) |
  ALT, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALT, Day 28 | 31.2 (28.37) | 27.5 (13.10) | 26.6 (8.02) | 33.7 (34.31)
  ALT, Day 35 | 25.0 (12.76) | 36.8 (31.13) | 23.8 (6.45) | 22.8 (9.33)
  ALT, Day 42 | 26.7 (20.29) | 27.8 (10.65) | 20.3 (8.36) | 21.2 (8.86)
  ALT, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALT, Day 49 | 19.4 (12.76) | 24.2 (12.19) | 18.5 (7.41) | 17.0 (6.10)
  ALT, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  ALT, Day 56 | 19.0 (9.49) | 21.2 (11.45) | 18.0 (6.14) | 14.7 (5.50)
  ALT, Day 63 | 15.2 (5.85) | 19.3 (7.69) | 18.4 (7.71) | 15.2 (2.64)
  AST, Baseline (Day 1) | 16.2 (2.99) | 19.2 (4.12) | 14.9 (3.14) | 17.8 (3.54)
  AST, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 2 | 14.8 (2.06) | 17.2 (2.64) |  | 17.5 (3.99)
  AST, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 3 | 15.5 (3.54) |  | 16.3 (2.25) |
  AST, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 5 | 18.8 (3.69) | 18.5 (4.14) |  | 15.7 (2.94)
  AST, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 6 | 15.0 (1.41) |  | 15.3 (3.01) |
  AST, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 7 | 19.8 (6.40) | 24.5 (10.88) |  | 16.0 (2.83)
  AST, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 8 | 15.0 (2.83) |  | 15.5 (2.14) |
  AST, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  AST, Day 11 | 17.0 (2.83) | 19.5 (3.11) |  | 13.8 (1.94)
  AST, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 12 | 16.5 (2.12) |  | 16.3 (3.33) |
  AST, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 14 | 24.8 (17.50) | 22.8 (6.55) |  | 15.7 (2.73)
  AST, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 15 | 16.0 (2.83) |  | 16.0 (3.59) |
  AST, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 21 | 17.0 (3.83) | 23.3 (5.79) |  | 18.8 (4.26)
  AST, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 22 | 17.5 (2.12) |  | 17.9 (2.47) |
  AST, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  AST, Day 28 | 23.6 (12.20) | 21.5 (5.13) | 21.9 (18.76) | 49.5 (80.64)
  AST, Day 35 | 20.0 (5.51) | 24.7 (10.03) | 19.5 (6.63) | 18.8 (5.19)
  AST, Day 42 | 21.5 (10.29) | 22.3 (2.66) | 15.9 (2.95) | 18.0 (3.35)
  AST, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  AST, Day 49 | 18.2 (4.97) | 19.5 (5.28) | 16.1 (5.41) | 16.5 (1.97)
  AST, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  AST, Day 56 | 18.0 (3.63) | 20.8 (4.09) | 16.9 (6.17) | 16.5 (2.17)
  AST, Day 63 | 15.2 (1.72) | 19.8 (6.34) | 16.1 (3.72) | 17.0 (3.41)

9. Primary Outcome: Part 3: Absolute Values of Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of bilirubin.
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 3 (Single Dose): VH4004280 450 mg Tablet
Number analyzed (Participants) | 6
μmol/L
  Direct Bilirubin, Baseline (Day 1) | 1.9950 (0.69810)
  Direct Bilirubin, Day 2 | 2.3085 (0.68186)
  Direct Bilirubin, Day 3 | 2.2515 (0.59646)
  Direct Bilirubin, Day 4 | 2.1660 (0.66375)
  Direct Bilirubin, Day 5 | 1.9380 (0.57905)
  Direct Bilirubin, Day 6 | 2.2800 (0.55848)
  Direct Bilirubin, Day 7 | 1.7670 (0.69810)
  Direct Bilirubin, Day 14 | 1.7385 (0.77549)
  Direct Bilirubin, Day 21 | 1.9380 (1.02979)
  Direct Bilirubin, Day 28 | 1.8525 (0.79043)
  Direct Bilirubin, Day 35 | 1.8525 (0.72077)
  Direct Bilirubin, Day 42: number analyzed (Participants) | 5
  Direct Bilirubin, Day 42 | 1.9494 (0.56196)
  Direct Bilirubin, Day 49 | 1.6530 (0.39981)
  Total Bilirubin, Baseline (Day 1) | 9.9750 (4.24640)
  Total Bilirubin, Day 2 | 12.2550 (4.31200)
  Total Bilirubin, Day 3 | 11.0580 (3.23487)
  Total Bilirubin, Day 4 | 10.4025 (2.63898)
  Total Bilirubin, Day 5 | 10.7730 (3.30875)
  Total Bilirubin, Day 6 | 11.3715 (2.69888)
  Total Bilirubin, Day 7 | 8.8635 (3.39669)
  Total Bilirubin, Day 14 | 8.7780 (5.31551)
  Total Bilirubin, Day 21 | 9.0915 (5.22647)
  Total Bilirubin, Day 28 | 8.8920 (4.03357)
  Total Bilirubin, Day 35 | 10.0890 (5.11859)
  Total Bilirubin, Day 42: number analyzed (Participants) | 5
  Total Bilirubin, Day 42 | 8.8920 (2.25240)
  Total Bilirubin, Day 49 | 8.4645 (2.29866)

10. Primary Outcome: Part 3: Absolute Values of Liver Panel Parameters: ALP, ALT and AST
Description: as for outcome 6
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 3 (Single Dose): VH4004280 450 mg Tablet
Number analyzed (Participants) | 6
IU/L
  ALP, Baseline (Day 1) | 55.7 (11.78)
  ALP, Day 2 | 47.8 (10.76)
  ALP, Day 3 | 50.2 (10.63)
  ALP, Day 4 | 50.8 (9.68)
  ALP, Day 5 | 48.8 (7.94)
  ALP, Day 6 | 49.7 (10.84)
  ALP, Day 7 | 50.3 (9.29)
  ALP, Day 14 | 60.2 (18.27)
  ALP, Day 21 | 58.0 (15.47)
  ALP, Day 28 | 59.7 (18.99)
  ALP, Day 35 | 59.5 (16.43)
  ALP, Day 42: number analyzed (Participants) | 5
  ALP, Day 42 | 58.2 (8.81)
  ALP, Day 49 | 55.8 (13.39)
  ALT, Baseline (Day 1) | 24.3 (17.07)
  ALT, Day 2 | 19.2 (13.04)
  ALT, Day 3 | 19.2 (11.00)
  ALT, Day 4 | 19.2 (8.80)
  ALT, Day 5 | 18.7 (8.36)
  ALT, Day 6 | 20.3 (9.20)
  ALT, Day 7 | 21.3 (10.78)
  ALT, Day 14 | 44.7 (64.91)
  ALT, Day 21 | 31.3 (34.51)
  ALT, Day 28 | 41.8 (57.78)
  ALT, Day 35 | 26.7 (22.90)
  ALT, Day 42: number analyzed (Participants) | 5
  ALT, Day 42 | 34.6 (47.24)
  ALT, Day 49 | 26.3 (30.80)
  AST, Baseline (Day 1) | 17.5 (4.28)
  AST, Day 2 | 15.2 (3.49)
  AST, Day 3 | 15.2 (3.37)
  AST, Day 4 | 15.7 (2.42)
  AST, Day 5 | 15.3 (2.80)
  AST, Day 6 | 17.5 (4.68)
  AST, Day 7 | 17.2 (5.23)
  AST, Day 14 | 24.3 (19.58)
  AST, Day 21 | 20.0 (7.97)
  AST, Day 28 | 24.5 (16.72)
  AST, Day 35 | 21.2 (7.91)
  AST, Day 42: number analyzed (Participants) | 5
  AST, Day 42 | 28.2 (27.31)
  AST, Day 49 | 19.5 (9.71)

11. Primary Outcome: Part 1: Change From Baseline in Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: Change from baseline was calculated by subtracting the baseline value from the post-dose visit value. Standard Deviation (SD)=0.0000 is defined as following: if all participants analyzed for a specific parameter at a specific time point have the same value, then SD is equal with 0.0000.
Time Frame: From Baseline (Day 1) and up to Day 49
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 10 | 6 | 7 | 6 | 6 | 6
μmol/L
  Direct Bilirubin, Baseline (Day 1) | 2.5650 (1.20915) | 1.9950 (0.69810) | 2.9314 (0.83439) | 2.2800 (1.39621) | 2.2800 (0.88304) | 2.8500 (0.88304)
  Direct Bilirubin, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  Direct Bilirubin, Day 2 | 0.0570 (0.80206) | 0.5130 (0.47141) | 0.0244 (0.96948) | -0.2280 (0.46726) | 0.4560 (0.69810) | 0.2280 (1.00100)
  Direct Bilirubin, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 3 | 0.1368 (0.87861) | 0.4845 (0.47656) | -0.1425 (0.62518) | -0.4275 (0.51584) | 0.0855 (0.57989) | 0.1995 (0.96379)
  Direct Bilirubin, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  Direct Bilirubin, Day 4 | -0.0684 (1.09107) | 0.0285 (0.39614) | -0.1140 (0.69810) | -0.4104 (0.84295) | -0.0285 (0.65264) | -0.1710 (0.85841)
  Direct Bilirubin, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 5 | 0.1710 (1.19564) | 0.6555 (0.36542) | -0.3420 (0.83072) | -0.3135 (0.62518) | 0.5415 (0.42464) | -0.0285 (0.58657)
  Direct Bilirubin, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 6 | 0.0000 (1.01004) | 0.6555 (0.45134) | -0.5415 (0.45134) | -0.4845 (0.54524) | 0.0855 (0.87695) | 0.0285 (0.95158)
  Direct Bilirubin, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 7 | 0.3249 (1.18869) | 0.4845 (0.60619) | -0.5700 (0.70643) | -0.3705 (0.67033) | 0.0570 (0.66375) | -0.2565 (0.69880)
  Direct Bilirubin, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  Direct Bilirubin, Day 14 | -0.2052 (1.04109) | -0.2850 (0.69810) | -1.1628 (1.04995) | -0.6555 (0.68755) | 0.1710 (0.72549) | -0.1710 (1.72023)
  Direct Bilirubin, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 21 | -0.0342 (1.03168) | 0.1425 (0.80509) | -0.5415 (0.86125) | -0.8550 (0.93034) | 0.1995 (0.55586) | -0.7980 (0.76218)
  Direct Bilirubin, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Direct Bilirubin, Day 28 | 0.2565 (1.37570) | 0.0855 (0.63753) | -0.4104 (0.44591) | -0.6270 (0.98331) | 0.9690 (0.60859) | -0.5130 (1.23310)
  Direct Bilirubin, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  Direct Bilirubin, Day 35 | -0.2052 (1.10174) | 0.1140 (0.27924) | -0.5700 (0.84928) | -0.5415 (1.02267) | 0.0000 (0.76474) | -0.7866 (0.67971)
  Direct Bilirubin, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Direct Bilirubin, Day 42 | 0.0855 (1.41321) |  |  | -0.6270 (0.84928) | 0.4560 (0.97134) | -0.0855 (0.77045)
  Direct Bilirubin, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Direct Bilirubin, Day 49 | 0.0855 (1.19333) |  |  | -0.7125 (0.96379) | 0.3705 (0.84756) | -0.1995 (0.95770)
  Total Bilirubin, Baseline (Day 1) | 13.1670 (6.84237) | 12.5400 (3.84908) | 14.9014 (3.65613) | 12.2550 (8.47558) | 11.6850 (5.00498) | 10.8300 (5.26132)
  Total Bilirubin, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  Total Bilirubin, Day 2 | 1.5770 (4.50462) | -0.6270 (1.14285) | -1.4657 (2.08465) | -1.4820 (1.96662) | 6.2985 (3.89252) | 5.4435 (4.21426)
  Total Bilirubin, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 3 | 1.1286 (4.54801) | -0.7695 (1.10159) | -2.9640 (1.07426) | -1.7955 (1.66407) | 3.8190 (4.03164) | 4.7595 (4.71342)
  Total Bilirubin, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 5
  Total Bilirubin, Day 4 | 0.4617 (5.19048) | -3.0780 (1.47100) | -0.8835 (3.77816) | -1.6416 (2.98785) | 4.1610 (2.59033) | 2.5650 (3.61332)
  Total Bilirubin, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 5 | 0.3933 (5.87628) | -0.8835 (0.97585) | -3.2775 (4.31980) | -1.5675 (2.78350) | 4.0470 (3.19851) | 3.9045 (2.63233)
  Total Bilirubin, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 6 | -0.2052 (6.38797) | -0.4275 (0.98973) | -5.4720 (3.74330) | -2.9070 (2.84087) | 2.2515 (4.45049) | 3.5340 (2.75234)
  Total Bilirubin, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 7 | 0.6840 (5.49629) | -1.9380 (1.87841) | -5.1585 (3.43777) | -1.5390 (2.91002) | 4.9875 (4.06738) | 1.7100 (3.37351)
  Total Bilirubin, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  Total Bilirubin, Day 14 | -2.7531 (6.09471) | -5.7855 (1.36978) | -6.7374 (3.07705) | -4.3035 (5.00001) | 1.1970 (2.11861) | 0.9690 (7.12039)
  Total Bilirubin, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 21 | -0.7353 (3.99004) | -2.9355 (2.88664) | -4.8165 (3.47667) | -4.7025 (5.15927) | 0.7980 (2.90532) | -1.9095 (4.55440)
  Total Bilirubin, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Total Bilirubin, Day 28 | 0.0000 (4.73683) | -3.4200 (1.69626) | -3.8304 (2.83984) | -4.2750 (5.88995) | 5.0730 (5.72446) | 0.5700 (6.01635)
  Total Bilirubin, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  Total Bilirubin, Day 35 | -1.1628 (4.21939) | -3.9615 (1.41183) | -5.0445 (4.68272) | -3.8190 (5.34403) | -0.3135 (3.91200) | -2.1888 (4.84024)
  Total Bilirubin, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Total Bilirubin, Day 42 | 0.0285 (5.67701) |  |  | -4.0470 (4.70877) | 3.9045 (5.91316) | 2.1375 (2.03985)
  Total Bilirubin, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  Total Bilirubin, Day 49 | -0.7695 (4.69270) |  |  | -3.4200 (4.88354) | 3.1350 (2.76717) | 1.9380 (8.15487)

12. Primary Outcome: Part 1: Change From Baseline in Liver Panel Parameters: ALP, ALT and AST
Description: Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.
Time Frame: From Baseline (Day 1) and up to Day 49
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 10 | 6 | 7 | 6 | 6 | 6
IU/L
  ALP, Baseline (Day 1) | 51.8 (9.39) | 64.7 (10.88) | 67.1 (27.91) | 69.0 (25.04) | 64.0 (11.10) | 61.8 (15.41)
  ALP, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  ALP, Day 2 | -4.2 (5.74) | -5.7 (2.88) | -6.7 (5.53) | -5.5 (5.09) | -5.8 (3.97) | -7.3 (7.23)
  ALP, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 3 | -3.6 (5.97) | -5.8 (3.97) | -9.5 (9.54) | -6.0 (6.20) | -8.2 (4.36) | -9.3 (6.47)
  ALP, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  ALP, Day 4 | -2.5 (6.19) | -4.2 (4.92) | -5.2 (12.46) | -5.4 (7.30) | -0.8 (2.86) | -9.0 (5.06)
  ALP, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 5 | -3.7 (3.47) | -5.5 (4.42) | -11.0 (10.33) | -5.7 (8.04) | -3.5 (3.62) | -4.2 (9.20)
  ALP, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 6 | -3.0 (4.92) | -2.2 (3.66) | -9.3 (11.66) | -6.0 (6.63) | -1.7 (2.80) | -7.3 (10.56)
  ALP, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 7 | -0.1 (6.95) | -0.3 (5.79) | -4.0 (14.86) | -4.7 (5.50) | 2.3 (4.23) | -5.0 (9.49)
  ALP, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  ALP, Day 14 | 3.0 (5.96) | -2.5 (5.61) | -6.8 (15.22) | -4.0 (5.18) | 2.0 (7.04) | -0.5 (8.29)
  ALP, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALP, Day 21 | 1.2 (3.49) | -6.0 (2.28) | -3.5 (6.80) | -3.0 (9.55) | -2.5 (4.59) | -2.7 (10.01)
  ALP, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  ALP, Day 28 | 2.1 (7.29) | -7.2 (7.33) | -0.2 (12.72) | -3.5 (5.89) | -0.5 (4.51) | 3.7 (17.44)
  ALP, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  ALP, Day 35 | 1.1 (4.07) | 1.7 (5.54) | -3.3 (6.83) | -5.2 (7.11) | 0.7 (7.20) | -0.6 (9.07)
  ALP, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  ALP, Day 42 | -1.8 (5.78) |  |  | -5.7 (3.67) | 2.2 (6.74) | 1.3 (6.44)
  ALP, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  ALP, Day 49 | -1.2 (4.45) |  |  | -1.8 (5.85) | 2.7 (9.35) | -2.2 (10.46)
  ALT, Baseline (Day 1) | 18.4 (5.60) | 22.8 (11.72) | 15.1 (4.85) | 20.7 (8.07) | 14.8 (2.93) | 16.0 (4.34)
  ALT, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  ALT, Day 2 | -0.1 (4.81) | -0.8 (5.64) | 0.4 (4.28) | 0.7 (1.75) | 0.8 (3.66) | -0.7 (1.86)
  ALT, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 3 | 0.2 (6.34) | -0.7 (6.44) | 1.5 (6.09) | 0.0 (1.26) | 1.0 (3.79) | 0.0 (1.79)
  ALT, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  ALT, Day 4 | 0.8 (7.13) | 0.3 (6.38) | 2.3 (7.37) | 2.6 (3.85) | -0.5 (3.73) | 0.2 (2.14)
  ALT, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 5 | -0.3 (7.97) | -1.2 (6.18) | 2.7 (9.37) | 3.8 (6.43) | 0.2 (2.93) | 0.0 (2.83)
  ALT, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 6 | 0.5 (9.57) | -0.3 (5.85) | 3.7 (11.29) | 3.5 (6.72) | -0.3 (3.98) | 2.8 (4.96)
  ALT, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 7 | 1.5 (11.65) | 0.7 (5.61) | 3.8 (10.87) | 4.0 (7.97) | 0.5 (4.51) | 4.8 (7.03)
  ALT, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  ALT, Day 14 | 7.7 (16.96) | 4.5 (11.26) | 5.2 (6.72) | 9.2 (14.58) | 6.2 (11.63) | 6.7 (10.03)
  ALT, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  ALT, Day 21 | 5.0 (14.54) | 0.7 (4.76) | 5.8 (8.42) | 3.8 (4.54) | 4.3 (5.16) | 6.2 (11.63)
  ALT, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  ALT, Day 28 | 1.7 (10.22) | 10.8 (20.21) | 4.8 (5.63) | 3.5 (4.09) | 2.0 (4.34) | 4.8 (6.88)
  ALT, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  ALT, Day 35 | 1.4 (9.88) | 5.7 (9.54) | 3.5 (4.76) | 2.8 (5.49) | 6.5 (15.36) | 2.4 (2.41)
  ALT, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  ALT, Day 42 | -1.7 (3.78) |  |  | 4.8 (7.70) | 1.5 (3.62) | 1.5 (2.74)
  ALT, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  ALT, Day 49 | -0.8 (2.64) |  |  | 7.2 (8.50) | 3.8 (9.75) | 1.2 (4.22)
  AST, Baseline (Day 1) | 17.3 (5.03) | 17.3 (5.82) | 15.1 (4.14) | 17.5 (3.62) | 15.0 (3.03) | 16.5 (3.51)
  AST, Day 2: number analyzed (Participants) | 9 | 6 | 7 | 6 | 6 | 6
  AST, Day 2 | -0.1 (3.69) | -1.0 (3.10) | -0.9 (4.34) | -1.0 (0.89) | 0.0 (3.29) | -0.7 (1.51)
  AST, Day 3: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 3 | -0.9 (3.25) | -1.3 (2.94) | 1.0 (3.69) | -0.8 (2.23) | -0.3 (2.50) | -1.3 (2.42)
  AST, Day 4: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  AST, Day 4 | -1.5 (3.95) | -0.7 (3.01) | 1.5 (2.81) | 1.0 (2.83) | -1.7 (2.07) | -1.0 (3.22)
  AST, Day 5: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 5 | -2.5 (4.48) | -2.5 (2.43) | 1.0 (3.22) | 1.0 (2.83) | -1.3 (2.07) | -0.7 (2.34)
  AST, Day 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 6 | -1.7 (5.12) | -1.3 (2.34) | 1.8 (4.92) | 0.2 (4.17) | -0.7 (2.50) | 0.2 (3.54)
  AST, Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 7 | -0.8 (5.87) | -0.5 (2.95) | 2.0 (3.22) | 0.7 (2.73) | 0.3 (1.63) | 1.5 (4.23)
  AST, Day 14: number analyzed (Participants) | 10 | 6 | 5 | 6 | 5 | 6
  AST, Day 14 | 22.7 (70.63) | 0.7 (3.50) | 0.6 (3.05) | 3.2 (5.12) | 4.6 (6.11) | 1.0 (1.79)
  AST, Day 21: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
  AST, Day 21 | 0.6 (7.37) | 1.3 (1.75) | 4.5 (6.35) | 2.0 (3.63) | 2.3 (3.01) | 1.7 (7.20)
  AST, Day 28: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  AST, Day 28 | -0.5 (4.88) | 5.7 (6.56) | 3.4 (3.97) | 2.8 (3.31) | 1.3 (3.27) | 0.3 (4.68)
  AST, Day 35: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
  AST, Day 35 | 0.1 (2.96) | 3.2 (5.31) | 4.5 (5.58) | 4.2 (5.34) | 3.5 (6.57) | 1.0 (1.58)
  AST, Day 42: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  AST, Day 42 | -1.0 (2.53) |  |  | 5.3 (4.72) | 1.3 (1.37) | 0.3 (3.61)
  AST, Day 49: number analyzed (Participants) | 6 | 0 | 0 | 6 | 6 | 6
  AST, Day 49 | -0.7 (1.75) |  |  | 5.8 (4.07) | 3.2 (4.71) | 1.5 (5.82)

13. Primary Outcome: Part 2: Change From Baseline in Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: as for outcome 11
Time Frame: From Baseline (Day 1) and up to Day 63
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 6 | 8 | 6
μmol/L
  Direct Bilirubin, Baseline (Day 1) | 2.2800 (0.88304) | 2.8500 (1.39621) | 2.1375 (0.79158) | 1.7100 (0.00000)
  Direct Bilirubin, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 2 | 0.0428 (0.84208) | 0.2565 (0.67323) |  | 0.4275 (0.40103)
  Direct Bilirubin, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 3 | -0.3420 (0.96732) |  | 0.0214 (0.51249) |
  Direct Bilirubin, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 5 | -0.0428 (1.13750) | 0.3135 (0.97585) |  | 0.4845 (0.54524)
  Direct Bilirubin, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 6 | -0.3420 (1.20915) |  | 0.2565 (0.78095) |
  Direct Bilirubin, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 7 | -0.2993 (1.01044) | 0.0570 (0.82837) |  | 0.8550 (0.47141)
  Direct Bilirubin, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 8 | -0.1710 (0.48366) |  | 0.3420 (0.69611) |
  Direct Bilirubin, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  Direct Bilirubin, Day 11 | 0.5130 (0.72549) | 0.5130 (0.60859) |  | 0.7695 (0.58989)
  Direct Bilirubin, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 12 | -0.5985 (1.81373) |  | 0.4061 (0.78062) |
  Direct Bilirubin, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 14 | -0.5558 (0.68932) | -0.2280 (0.95923) |  | 0.2850 (0.33625)
  Direct Bilirubin, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 15 | 0.1710 (0.96732) |  | 0.7481 (0.46551) |
  Direct Bilirubin, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 21 | -0.4275 (0.86632) | -0.1140 (1.00100) |  | 0.8835 (0.34905)
  Direct Bilirubin, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 22 | 0.9405 (1.08824) |  | 1.0901 (0.85225) |
  Direct Bilirubin, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  Direct Bilirubin, Day 28 | -0.8208 (1.13041) | -0.8265 (0.87472) | -0.0428 (0.67632) | 0.1710 (0.49561)
  Direct Bilirubin, Day 35 | -0.4845 (0.79043) | -0.9690 (0.91556) | 0.0000 (0.80725) | 0.0855 (0.41536)
  Direct Bilirubin, Day 42 | -0.2280 (0.54791) | -0.7695 (0.80024) | -0.1069 (1.08896) | -0.1140 (0.35322)
  Direct Bilirubin, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  Direct Bilirubin, Day 49 | -0.2736 (0.35459) | -0.6270 (0.84928) | 0.0641 (0.45645) | 0.1995 (0.59646)
  Direct Bilirubin, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  Direct Bilirubin, Day 56 | -0.3705 (0.83364) | -0.7866 (0.82542) | -0.2565 (0.62663) | 0.0855 (0.49265)
  Direct Bilirubin, Day 63 | -0.5130 (0.64890) | -0.9405 (1.25542) | -0.2779 (0.80174) | 0.2565 (0.51584)
  Total Bilirubin, Baseline (Day 1) | 11.9700 (3.42000) | 15.1050 (6.87553) | 9.6188 (3.53265) | 8.2650 (1.28724)
  Total Bilirubin, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 2 | -0.0855 (2.38789) | 2.8500 (3.18017) |  | 3.3915 (2.22541)
  Total Bilirubin, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 3 | 1.7955 (0.36275) |  | 2.5864 (2.03655) |
  Total Bilirubin, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 5 | -0.0855 (2.68748) | 3.7620 (4.99952) |  | 4.8165 (3.79823)
  Total Bilirubin, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 6 | 0.5985 (1.33007) |  | 3.6338 (2.33168) |
  Total Bilirubin, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 7 | -1.6673 (1.34192) | 1.3965 (4.31166) |  | 6.6120 (2.54018)
  Total Bilirubin, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 8 | 2.0520 (2.90197) |  | 4.8094 (3.07316) |
  Total Bilirubin, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  Total Bilirubin, Day 11 | -0.8550 (3.62746) | 3.6765 (2.12893) |  | 4.7880 (1.89494)
  Total Bilirubin, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 12 | -3.0780 (6.77125) |  | 6.0705 (2.04180) |
  Total Bilirubin, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 14 | -3.2918 (0.94050) | -0.8550 (5.47307) |  | 5.7000 (1.55099)
  Total Bilirubin, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 15 | 1.0260 (1.93464) |  | 5.3651 (2.82455) |
  Total Bilirubin, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 21 | -3.0780 (1.45769) | 0.7125 (4.72334) |  | 6.6975 (1.87139)
  Total Bilirubin, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 22 | 5.3865 (0.12092) |  | 8.4645 (4.99216) |
  Total Bilirubin, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  Total Bilirubin, Day 28 | -4.0014 (3.67869) | -4.7880 (6.47907) | 0.1069 (3.43820) | 1.5105 (3.13339)
  Total Bilirubin, Day 35 | -2.6790 (2.91336) | -4.3320 (5.66489) | 0.6840 (1.99837) | 0.8550 (1.00294)
  Total Bilirubin, Day 42 | -1.3395 (1.08913) | -4.3605 (5.70510) | 0.5985 (4.89669) | 0.6270 (2.71598)
  Total Bilirubin, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  Total Bilirubin, Day 49 | -0.7866 (1.70400) | -2.9640 (4.81803) | 1.5604 (2.81789) | 1.5105 (2.40233)
  Total Bilirubin, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  Total Bilirubin, Day 56 | -1.8525 (2.73047) | -6.0534 (4.17394) | -1.3039 (2.45421) | 0.5415 (1.86199)
  Total Bilirubin, Day 63 | -3.0495 (1.72504) | -4.7595 (5.86150) | -0.6413 (2.44536) | 1.9095 (2.35811)

14. Primary Outcome: Part 2: Change From Baseline in Liver Panel Parameters: ALP, ALT and AST
Description: Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.
Time Frame: From Baseline (Day 1) and up to Day 63
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 6 | 8 | 6
IU/L
  ALP, Baseline (Day 1) | 66.2 (16.75) | 53.7 (10.01) | 57.5 (21.37) | 56.7 (11.41)
  ALP, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 2 | 4.0 (8.45) | -1.7 (3.33) |  | -0.5 (2.81)
  ALP, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 3 | -0.5 (4.95) |  | 0.9 (3.31) |
  ALP, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 5 | -0.8 (4.50) | -3.8 (5.98) |  | 0.5 (4.85)
  ALP, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 6 | -4.5 (3.54) |  | -1.9 (3.40) |
  ALP, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 7 | -0.3 (5.56) | -4.8 (7.47) |  | -0.2 (5.27)
  ALP, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 8 | 0.0 (8.49) |  | -1.8 (3.77) |
  ALP, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  ALP, Day 11 | -7.5 (3.54) | -2.0 (5.48) |  | -2.3 (5.05)
  ALP, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 12 | 2.5 (4.95) |  | 0.8 (3.24) |
  ALP, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 14 | 4.5 (14.57) | -6.0 (6.16) |  | 1.3 (4.37)
  ALP, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 15 | -2.5 (6.36) |  | 0.5 (4.99) |
  ALP, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 21 | -3.0 (3.16) | -3.2 (9.02) |  | 0.8 (4.62)
  ALP, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 22 | 2.0 (5.66) |  | 5.1 (3.94) |
  ALP, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALP, Day 28 | -2.0 (4.85) | -4.5 (6.69) | 2.3 (5.70) | 2.8 (3.76)
  ALP, Day 35 | -2.0 (5.83) | -0.7 (8.62) | 2.4 (7.41) | -3.7 (3.61)
  ALP, Day 42 | 1.5 (6.47) | -2.3 (5.43) | 4.6 (9.64) | 1.0 (4.73)
  ALP, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALP, Day 49 | 0.8 (7.89) | -2.7 (7.03) | 1.3 (6.76) | -2.7 (4.55)
  ALP, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  ALP, Day 56 | 2.8 (9.20) | -3.6 (3.21) | 5.3 (6.90) | -0.2 (4.96)
  ALP, Day 63 | 0.3 (5.05) | 0.2 (5.95) | 1.3 (4.37) | 0.7 (2.88)
  ALT, Baseline (Day 1) | 18.7 (11.98) | 19.0 (6.93) | 16.3 (5.04) | 19.5 (7.69)
  ALT, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 2 | -1.5 (5.80) | 0.2 (2.64) |  | 0.3 (2.07)
  ALT, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 3 | -2.0 (1.41) |  | 2.0 (2.33) |
  ALT, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 5 | 1.5 (8.96) | 0.5 (3.83) |  | -2.8 (2.64)
  ALT, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 6 | -6.0 (4.24) |  | 2.0 (5.45) |
  ALT, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 7 | 4.8 (8.38) | 5.7 (7.81) |  | -3.0 (3.79)
  ALT, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 8 | -6.0 (2.83) |  | 0.5 (6.02) |
  ALT, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  ALT, Day 11 | 9.0 (5.66) | 4.0 (11.28) |  | -4.7 (4.72)
  ALT, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 12 | -2.0 (1.41) |  | 2.9 (9.48) |
  ALT, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 14 | 15.8 (17.21) | 10.5 (13.85) |  | -2.8 (5.53)
  ALT, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 15 | -1.0 (2.83) |  | 5.3 (10.74) |
  ALT, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 21 | 7.0 (4.69) | 13.8 (15.28) |  | 3.7 (9.48)
  ALT, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 22 | 0.5 (6.36) |  | 7.9 (10.29) |
  ALT, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALT, Day 28 | 12.0 (15.98) | 8.5 (9.65) | 10.4 (9.38) | 14.2 (37.02)
  ALT, Day 35 | 6.3 (5.50) | 17.8 (26.69) | 7.5 (7.29) | 3.3 (12.23)
  ALT, Day 42 | 8.0 (8.65) | 8.8 (7.19) | 4.0 (6.74) | 1.7 (8.07)
  ALT, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALT, Day 49 | 0.2 (1.10) | 5.2 (7.60) | 2.3 (6.34) | -2.5 (5.96)
  ALT, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  ALT, Day 56 | 0.3 (3.33) | 0.8 (8.44) | 1.8 (6.71) | -4.8 (2.48)
  ALT, Day 63 | -3.5 (6.53) | 0.3 (3.88) | 2.1 (6.31) | -4.3 (5.92)
  AST, Baseline (Day 1) | 16.2 (2.99) | 19.2 (4.12) | 14.9 (3.14) | 17.8 (3.54)
  AST, Day 2: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 2 | -1.3 (2.06) | -2.0 (2.68) |  | -0.3 (1.51)
  AST, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 3 | -1.0 (1.41) |  | 1.4 (3.02) |
  AST, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 5 | 2.8 (3.86) | -0.7 (3.50) |  | -2.2 (2.04)
  AST, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 6 | -1.5 (0.71) |  | 0.4 (3.89) |
  AST, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 7 | 3.8 (4.11) | 5.3 (9.73) |  | -1.8 (3.06)
  AST, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 8 | -1.5 (0.71) |  | 0.6 (2.88) |
  AST, Day 11: number analyzed (Participants) | 2 | 4 | 0 | 6
  AST, Day 11 | 2.0 (1.41) | 2.0 (6.06) |  | -4.0 (2.53)
  AST, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 12 | 0.0 (0.00) |  | 1.4 (4.44) |
  AST, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 14 | 8.8 (14.36) | 3.7 (6.35) |  | -2.2 (2.93)
  AST, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 15 | -0.5 (0.71) |  | 1.1 (4.79) |
  AST, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 21 | 1.0 (1.15) | 4.2 (5.81) |  | 1.0 (3.10)
  AST, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 22 | 1.0 (0.00) |  | 3.0 (3.02) |
  AST, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  AST, Day 28 | 7.8 (9.31) | 2.3 (6.22) | 7.0 (17.57) | 31.7 (81.01)
  AST, Day 35 | 3.8 (4.67) | 5.5 (7.29) | 4.6 (5.68) | 1.0 (6.42)
  AST, Day 42 | 5.3 (7.71) | 3.2 (5.27) | 1.0 (2.27) | 0.2 (3.87)
  AST, Day 49: number analyzed (Participants) | 5 | 6 | 8 | 6
  AST, Day 49 | 2.4 (2.41) | 0.3 (4.03) | 1.3 (3.20) | -1.3 (4.13)
  AST, Day 56: number analyzed (Participants) | 6 | 5 | 8 | 6
  AST, Day 56 | 1.8 (2.64) | 0.4 (3.85) | 2.0 (7.46) | -1.3 (1.63)
  AST, Day 63 | -1.0 (1.41) | 0.7 (4.03) | 1.3 (4.30) | -0.8 (3.54)

15. Primary Outcome: Part 3: Change From Baseline in Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.
Time Frame: From Baseline (Day 1) and up to Day 49
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 3 (Single Dose): VH4004280 450 mg Tablet
Number analyzed (Participants) | 6
μmol/L
  Direct Bilirubin, Baseline (Day 1) | 1.9950 (0.69810)
  Direct Bilirubin, Day 2 | 0.3135 (0.43820)
  Direct Bilirubin, Day 3 | 0.2565 (0.40103)
  Direct Bilirubin, Day 4 | 0.1710 (0.55146)
  Direct Bilirubin, Day 5 | -0.0570 (0.62752)
  Direct Bilirubin, Day 6 | 0.2850 (0.50341)
  Direct Bilirubin, Day 7 | -0.2280 (0.65488)
  Direct Bilirubin, Day 14 | -0.2565 (0.23571)
  Direct Bilirubin, Day 21 | -0.0570 (0.54791)
  Direct Bilirubin, Day 28 | -0.1425 (0.39614)
  Direct Bilirubin, Day 35 | -0.1425 (0.22729)
  Direct Bilirubin, Day 42: number analyzed (Participants) | 5
  Direct Bilirubin, Day 42 | -0.1026 (0.72145)
  Direct Bilirubin, Day 49 | -0.3420 (0.50727)
  Total Bilirubin, Baseline (Day 1) | 9.9750 (4.24640)
  Total Bilirubin, Day 2 | 2.2800 (1.65673)
  Total Bilirubin, Day 3 | 1.0830 (2.10730)
  Total Bilirubin, Day 4 | 0.4275 (2.53346)
  Total Bilirubin, Day 5 | 0.7980 (2.64396)
  Total Bilirubin, Day 6 | 1.3965 (2.58072)
  Total Bilirubin, Day 7 | -1.1115 (3.11530)
  Total Bilirubin, Day 14 | -1.1970 (2.45193)
  Total Bilirubin, Day 21 | -0.8835 (2.28249)
  Total Bilirubin, Day 28 | -1.0830 (2.22344)
  Total Bilirubin, Day 35 | 0.1140 (3.42285)
  Total Bilirubin, Day 42: number analyzed (Participants) | 5
  Total Bilirubin, Day 42 | -2.0520 (4.26987)
  Total Bilirubin, Day 49 | -1.5105 (2.99795)

16. Primary Outcome: Part 3: Change From Baseline in Liver Panel Parameters: ALP, ALT and AST
Description: Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.
Time Frame: From Baseline (Day 1) and up to Day 49
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 3 (Single Dose): VH4004280 450 mg Tablet
Number analyzed (Participants) | 6
IU/L
  ALP, Baseline (Day 1) | 55.7 (11.78)
  ALP, Day 2 | -7.8 (3.13)
  ALP, Day 3 | -5.5 (3.02)
  ALP, Day 4 | -4.8 (2.86)
  ALP, Day 5 | -6.8 (5.64)
  ALP, Day 6 | -6.0 (2.61)
  ALP, Day 7 | -5.3 (4.89)
  ALP, Day 14 | 4.5 (9.81)
  ALP, Day 21 | 2.3 (9.87)
  ALP, Day 28 | 4.0 (12.20)
  ALP, Day 35 | 3.8 (8.16)
  ALP, Day 42: number analyzed (Participants) | 5
  ALP, Day 42 | -0.2 (5.93)
  ALP, Day 49 | 0.2 (6.05)
  ALT, Baseline (Day 1) | 24.3 (17.07)
  ALT, Day 2 | -5.2 (4.49)
  ALT, Day 3 | -5.2 (6.40)
  ALT, Day 4 | -5.2 (8.57)
  ALT, Day 5 | -5.7 (8.87)
  ALT, Day 6 | -4.0 (8.44)
  ALT, Day 7 | -3.0 (7.32)
  ALT, Day 14 | 20.3 (48.50)
  ALT, Day 21 | 7.0 (17.85)
  ALT, Day 28 | 17.5 (41.15)
  ALT, Day 35 | 2.3 (6.53)
  ALT, Day 42: number analyzed (Participants) | 5
  ALT, Day 42 | 10.2 (28.44)
  ALT, Day 49 | 2.0 (15.07)
  AST, Baseline (Day 1) | 17.5 (4.28)
  AST, Day 2 | -2.3 (2.58)
  AST, Day 3 | -2.3 (3.33)
  AST, Day 4 | -1.8 (3.13)
  AST, Day 5 | -2.2 (2.79)
  AST, Day 6 | 0.0 (3.63)
  AST, Day 7 | -0.3 (3.08)
  AST, Day 14 | 6.8 (15.46)
  AST, Day 21 | 2.5 (4.04)
  AST, Day 28 | 7.0 (12.59)
  AST, Day 35 | 3.7 (6.35)
  AST, Day 42: number analyzed (Participants) | 5
  AST, Day 42 | 10.6 (22.61)
  AST, Day 49 | 2.0 (6.87)

17. Primary Outcome: Part 1: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Parameters
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of the liver panel parameters: ALT, ALP, AST, total bilirubin and direct bilirubin. The number of participants with any grade increase (from grade 1 [mild] to grade 4 [potentially life-threatening]) have been presented.
Time Frame: Up to Day 49
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 10 | 6 | 7 | 6 | 6 | 6
Participants
  ALT, Increase to Grade 1 | 1 | 1 | 0 | 1 | 0 | 0
  ALT, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Increase to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Increase to Grade 3 | 1 | 0 | 0 | 0 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0 | 1 | 0
  Total Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Part 2: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Parameters
Description: as for outcome 17
Time Frame: Up to Day 63
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 6 | 8 | 6
Participants
  ALT, Increase to Grade 1 | 1 | 1 | 0 | 1
  ALT, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 1 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0 | 0 | 0
  AST, Increase to Grade 1 | 1 | 0 | 1 | 0
  AST, Increase to Grade 2 | 0 | 0 | 0 | 0
  AST, Increase to Grade 3 | 0 | 0 | 0 | 1
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0

19. Primary Outcome: Part 3: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Parameters
Description: as for outcome 17
Time Frame: Up to Day 49
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 (Single Dose): VH4004280 450 mg Tablet
Number analyzed (Participants) | 6
Participants
  ALT, Increase to Grade 1 | 0
  ALT, Increase to Grade 2 | 1
  ALT, Increase to Grade 3 | 0
  ALT, Increase to Grade 4 | 0
  ALP, Increase to Grade 1 | 0
  ALP, Increase to Grade 2 | 0
  ALP, Increase to Grade 3 | 0
  ALP, Increase to Grade 4 | 0
  AST, Increase to Grade 1 | 1
  AST, Increase to Grade 2 | 0
  AST, Increase to Grade 3 | 0
  AST, Increase to Grade 4 | 0
  Total Bilirubin, Increase to Grade 1 | 0
  Total Bilirubin, Increase to Grade 2 | 0
  Total Bilirubin, Increase to Grade 3 | 0
  Total Bilirubin, Increase to Grade 4 | 0
  Direct Bilirubin, Increase to Grade 1 | 0
  Direct Bilirubin, Increase to Grade 2 | 0
  Direct Bilirubin, Increase to Grade 3 | 0
  Direct Bilirubin, Increase to Grade 4 | 0

20. Primary Outcome: Part 1: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC[0-infinity]) Following Single Dose Administration of VH4004280
Description: Blood samples were collected as assessed by protocol, at specific time points for pharmacokinetic (PK) analysis to determine AUC(0-inf). For AUC, a linear trapezoidal method was employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method was used for those arising from decreasing concentrations. Geometric Coefficient of Variation was expressed in percentages.
Time Frame: At Day 1
Population: The analysis was performed on the VH4004280 PK Set which included all participants in the Part 1 (SAD) Safety Set who received 1 full dose of study treatment with at least one non-missing PK assessment. The participants were analyzed according to the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
Hour nanogram per milliliter (h*ng/mL) | 1396.25 (28.02) | 16829.76 (17.59) | 51168.22 (51.76) | 174441.72 (33.21) | 215339.87 (42.90)

21. Primary Outcome: Part 2: AUC Over a Dosing Interval From Time of Dosing to the Time of the Subsequent Dose (AUC[0-t]) Following Repeat Dose Administration of VH4004280
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine AUC(0-t). For AUC, a linear trapezoidal method was employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method was used for those arising from decreasing concentrations.
Time Frame: At Days 1 and 14 for Part 2 (MAD): VH4004280 100 mg PiB and Part 2 (MAD): VH4004280 350 mg PiB groups, and at Days 2 and 15 for Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB group
Population: The analysis was performed on the VH4004280 PK Set which included all participants in the Part 2 (MAD) Safety Set who received at least 1 full dose of study treatment with at least one non-missing PK assessment. The participants were analyzed according to the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 8 | 6
h*ng/mL
  Day 1: number analyzed (Participants) | 6 | 0 | 6
  Day 1 | 6268.14 (17.35) |  | 14869.75 (23.49)
  Day 2: number analyzed (Participants) | 0 | 8 | 0
  Day 2 |  | 15157.94 (26.00) |
  Day 14: number analyzed (Participants) | 6 | 0 | 6
  Day 14 | 449239.54 (53.50) |  | 1882862.73 (37.66)
  Day 15: number analyzed (Participants) | 0 | 8 | 0
  Day 15 |  | 1527149.1 (26.00) |

22. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) Following Single Dose Administration of VH4004280
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine Cmax.
Time Frame: At Day 1
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 13.49 (23.59) | 149.77 (27.34) | 438.80 (53.60) | 1342.72 (30.74) | 1630.95 (27.05)

23. Primary Outcome: Part 1: Time to Maximum Observed Plasma Concentration (Tmax) Following Single Dose Administration of VH4004280
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine Tmax.
Time Frame: At Day 1
Population: The analysis was performed on the VH4004280 PK Set which included all participants in the Part 1 (SAD) Safety Set who received at least 1 full dose of study treatment with at least one non-missing PK assessment. The participants were analyzed according to the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
hours | 9.63 (9.13) | 9.90 (16.62) | 11.15 (40.09) | 10.31 (7.45) | 8.53 (20.71)

24. Primary Outcome: Part 1: Apparent Terminal Half-life (T1/2) Following Single Dose Administration of VH4004280
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine T1/2.
Time Frame: Day 1 to Day 49
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
hours | 145.82 (40.60) | 149.91 (40.40) | 149.94 (43.47) | 177.58 (18.23) | 172.66 (29.45)

25. Primary Outcome: Part 2: Cmax Following Repeat Dose Administration of VH4004280
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine Cmax.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 8 | 6
ng/mL
  Day 1: number analyzed (Participants) | 6 | 0 | 6
  Day 1 | 422.68 (15.53) |  | 957.92 (21.70)
  Day 2: number analyzed (Participants) | 0 | 8 | 0
  Day 2 |  | 972.51 (26.49) |
  Day 14: number analyzed (Participants) | 6 | 0 | 6
  Day 14 | 1725.63 (36.64) |  | 7573.63 (66.10)
  Day 15: number analyzed (Participants) | 0 | 8 | 0
  Day 15 |  | 4487.14 (42.27) |

26. Primary Outcome: Part 2: T1/2 Following Repeat Dose Administration of VH4004280
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine T1/2.
Time Frame: Day 14 to Day 63 for Part 2 (MAD): VH4004280 100 mg PiB and Part 2 (MAD): VH4004280 350 mg PiB groups, and Day 15 to Day 63 for Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB group
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 8 | 6
hours
  Day 14 to Day 63: number analyzed (Participants) | 6 | 0 | 6
  Day 14 to Day 63 | 166.29 (34.95) |  | 147.93 (56.42)
  Day 15 to Day 63: number analyzed (Participants) | 0 | 8 | 0
  Day 15 to Day 63 |  | 207.76 (35.36) |

27. Primary Outcome: Part 2: Tmax Following Repeat Dose Administration of VH4004280
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine Tmax.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB
Number analyzed (Participants) | 6 | 8 | 6
hours
  Day 1: number analyzed (Participants) | 6 | 0 | 6
  Day 1 | 9.28 (11.56) |  | 9.57 (15.66)
  Day 2: number analyzed (Participants) | 0 | 8 | 0
  Day 2 |  | 9.68 (13.38) |
  Day 14: number analyzed (Participants) | 6 | 0 | 6
  Day 14 | 9.58 (15.72) |  | 15.49 (50.84)
  Day 15: number analyzed (Participants) | 0 | 8 | 0
  Day 15 |  | 9.33 (21.14) |

ADVERSE EVENTS:
Time Frame: All cause mortality, serious adverse events (SAEs) and non-SAEs were collected up to a 49-day period following VH4004280 or placebo (i.e.: Day 49 for Parts 1 and 3, and Day 63 for Part 2).
Description: The analysis was performed on the Safety Set which included all participants who received at least 1 full or partial dose of study treatment.
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) | Part 1 (SAD): VH4004280 10 mg PiB | Part 1 (SAD): VH4004280 50 mg PiB | Part 1 (SAD): VH4004280 150 mg PiB | Part 1 (SAD): VH4004280 450 mg PiB | Part 1 (SAD): VH4004280 900 mg PiB | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4004280 100 mg PiB | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4004280 350 mg PiB | Part 3 (Single Dose): VH4004280 450 mg Tablet
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/10 | 2/6 | 3/7 | 0/6 | 0/6 | 1/6 | 3/6 | 4/6 | 7/8 | 4/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-bottle (PiB) (N=10) | Part 1 (SAD): VH4004280 10 mg PiB (N=6) | Part 1 (SAD): VH4004280 50 mg PiB (N=7) | Part 1 (SAD): VH4004280 150 mg PiB (N=6) | Part 1 (SAD): VH4004280 450 mg PiB (N=6) | Part 1 (SAD): VH4004280 900 mg PiB (N=6) | Part 2 Multiple Ascending Dose (MAD): Placebo PiB (N=6) | Part 2 (MAD): VH4004280 100 mg PiB (N=6) | Part 2 (MAD): VH4004280 250 mg + Midazolam (MDZ) PiB (N=8) | Part 2 (MAD): VH4004280 350 mg PiB (N=6) | Part 3 (Single Dose): VH4004280 450 mg Tablet (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bile acids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT05163522/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT05163522/SAP_001.pdf